CLINICAL TRIAL: NCT01725880
Title: Long-term Follow-up (LTFU) Study of the Phase I/II Safety and Preliminary Efficacy Investigation of Intramedullary Spinal Cord Transplantation of HuCNS-SC® in Subjects With Thoracic (T2-T11) Spinal Cord Trauma
Brief Title: Long-Term Follow-Up of Transplanted Human Central Nervous System Stem Cells (HuCNS-SC) in Spinal Cord Trauma Subjects
Status: Terminated | Type: Observational
Why Stopped: Based on a business decision unrelated to any safety concerns.
Sponsor: StemCells, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CL-N03-SC; TpP_I_2012_002 (Other: SwissMedic)
Record Dates: First submitted 2012-11-09; First posted 2012-11-14 (Estimated); Last update posted 2016-06-03 (Estimated); Status verified 2016-05

CONDITIONS: Spinal Cord Injury
Keywords: Spinal Cord Injury; HuCNS-SC cells; Human Neural Stem Cells; Neural Stem Cells; Stem Cells
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- No treatment: Observation
  Interventions: Other: Observation

INTERVENTIONS:
Other: Observation

SUMMARY:
The purpose of this study is to determine the long term safety and preliminary efficacy of intramedullary transplantation of HuCNS-SC cells in subjects with thoracic spinal cord trauma.

DETAILED DESCRIPTION:
The investigation is a multi-year observational study following the completion of the open-label, single dose Phase I/II study involving transplantation of allogeneic HuCNS-SC cells into 12 subjects with thoracic spinal cord injury.

Subjects will be monitored at routine intervals for safety and preliminary efficacy for four years. The LTFU study will commence following the one year post-transplantation termination visit of the Phase I/II investigation.

ELIGIBILITY:
Inclusion Criteria:

* Must have undergone HuCNS-SC transplantation as a subject in the Phase I/II trial
* Must agree to comply in good faith with all conditions of the study and to attend all required study visits

Exclusion Criteria:

* Subjects have received or are receiving off-protocol immunosuppressive medications
* Subjects who, after completion of Phase I/II trial (Protocol # CL-N02-SC), have entered or are about to enter any other investigational study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who had undergone intramedullary transplantation of HuCNS-SC cells in the thoracic region.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2012-11; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
American Spinal Injury Association (ASIA) Impairment Scale Improvement | Four years
  Evidence of improvement in ASIA impairment scale as confirmed by neurological examination

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Huhn, M.D., Study Director — StemCells, Inc.
Locations (1):
- Uniklinik Balgrist, Zurich, Switzerland

REFERENCES:
- See also: Spinal Cord Injury Trial — http://www.stemcellsinc.com/Therapeutic-Programs/Spinal-Cord-Injury.htm